CLINICAL TRIAL: NCT02143128
Title: Safety and Quality for Inpatients After Surgery at the Ward. Development and Evaluation of a New Tool: Efficacy Side-effect Score (ESS)
Brief Title: Efficacy Side-effect Score (ESS): Development and Evaluation of a New Tool for Patients After Surgery
Acronym: ESScore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre VikenHF Kongsberg Sykehus (Other)
Collaborators: Norwegian Medical Association (Other)
Responsible Party: Principal Investigator, Erlend Johan Skraastad, Consultant, MD, Vestre VikenHF Kongsberg Sykehus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VVHF-KS001
Record Dates: First submitted 2014-05-14; First posted 2014-05-20 (Estimated); Results first posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Pain; Postoperative Vomiting and Nausea; Postoperative Complications; Mental Status Changes Postoperative
Keywords: score; postoperative; pain; nausea; mental status; tool
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Postoperative Complications; Pain; Nausea

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Efficacy Safety Score (Experimental): Patients assessed using the ESS
  Interventions: Other: Efficacy Safety Score
- Verbal Numeric Rating Scale (Active Comparator): Patients assessed using VNRS
  Interventions: Other: Verbal Numeric Rating Scale
- Control (No Intervention): Regular follow up

INTERVENTIONS:
Other: Efficacy Safety Score — Evaluation using the score for postoperative patients
  Other Names: ESS
  Arms: Efficacy Safety Score
Other: Verbal Numeric Rating Scale — Patients assessed for postoperative pain using VNRS (0-10)
  Other Names: VNRS
  Arms: Verbal Numeric Rating Scale

SUMMARY:
We hypothesized that better control of postoperative pain treatment and its side effects by monitoring ESS might influence the degree of mobility and morbidity in surgical patients and consequently reduce LOS. Thus, our aim was to validate the influence of recording ESS and the application of a "call-out algorithm" on LOS in two university hospitals in which the routine policy of registration of pain had not been adopted yet.

DETAILED DESCRIPTION:
Using clinical experience and consensus-methodology the investigators picked up and digitalized information about mental, postoperative nausea, vomiting and pain status at the rest and during mobilization in so called Efficacy Safety Score (ESS). Depending on expression of patient's complaints, all mentioned above clinical features are scored. We hypothesized that better control of postoperative pain treatment and its side effects by monitoring ESS might influence the degree of mobility and morbidity in surgical patients and consequently reduce length of hospital stay (LOS). Thus, our aim was to validate the influence of recording ESS and the application of a "call-out algorithm" on LOS in two university hospitals in which the routine policy of registration of pain had not been adopted yet. The primary endpoint of the study was to assess LOS in groups of patients with different types of clinical data records and "call-out algorithms," while secondary endpoints were to compare the degree of mobilization, number of postoperative nonsurgical complications, and 28-day survival between the groups.and summarized in the total score.

ELIGIBILITY:
Inclusion Criteria:

* All adult postoperative patients that are inpatients, and scheduled for hospitalization for more than 8 hours

Exclusion Criteria:

* Children, mental illness, communication difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1152 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Kuklin, Dr med, Principal Investigator — Vestre VIkenHF, Kongsberg
Locations (2):
- Astana University Hospital, Astana, Astana, Kazakhstan
- Krasnodar University Hospital, Krasnodar, Russia

IPD SHARING:
Plan to Share IPD: Yes
On reasonable request
Supporting Information: SAP, CSR, Analytic Code
Time Frame: After end of study
Access Criteria: Contact PI, Vladimir Kuklin
URL: https://doi.org/10.1155/2017/9431984

REFERENCES:
- [Derived] Dybvik L, Skraastad E, Yeltayeva A, Konkayev A, Musaeva T, Zabolotskikh I, Bjertnaes L, Dahl V, Raeder J, Kuklin V. Influence of a New "Call-Out Algorithm" for Management of Postoperative Pain and Its Side Effects on Length of Stay in Hospital: A Two-Centre Prospective Randomized Trial. Pain Res Manag. 2017;2017:9431984. doi: 10.1155/2017/9431984. Epub 2017 Aug 10. PMID 28855800

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Efficacy Safety Score | Verbal Numeric Rating Scale | Control
Started | 409 | 417 | 326
Completed | 409 | 417 | 326
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efficacy Safety Score | Verbal Numeric Rating Scale | Control | Total
Number analyzed (Participants) | 409 | 417 | 326 | 1152
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Different sites contributing to total.
  years
    Astana: number analyzed (Participants) | 228 | 227 | 224 | 679
    Astana | 43.4 (16.4) | 42.4 (16.4) | 44.9 (15.8) | 43.6 (16.2)
    Krasnodar: number analyzed (Participants) | 181 | 190 | 102 | 473
    Krasnodar | 55.2 (14.7) | 55.1 (15.6) | 56 (14.9) | 55.4 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Overall number constitutes of number analyzed at two locations.
  Participants
    Kazakhstan, Astana: number analyzed (Participants) | 228 | 227 | 224 | 679
    Kazakhstan, Astana: Female | 112 | 95 | 104 | 311
    Kazakhstan, Astana: Male | 116 | 132 | 120 | 368
    Russia, Krasnodar: number analyzed (Participants) | 181 | 190 | 102 | 473
    Russia, Krasnodar: Female | 112 | 121 | 53 | 286
    Russia, Krasnodar: Male | 69 | 69 | 49 | 187
Region of Enrollment [Number; unit: participants]
  Kazakhstan | 228 | 227 | 224 | 679
  Russia | 181 | 190 | 102 | 473

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay (LOS)
Description: Assess LOS in groups of patients with different types of clinical data records an "all-out algorithms"
Time Frame: 28 days
Measure: Mean (Full Range); unit: days
Arm/Group | Efficacy Safety Score | Verbal Numeric Rating Scale | Control
Number analyzed (Participants) | 409 | 417 | 326
days | 12.7 [6.4 to 19.0] | 13.5 [7.3 to 19.7] | 14.2 [8.0 to 20.4]

ADVERSE EVENTS:
Arm/Group | Efficacy Safety Score | Verbal Numeric Rating Scale | Control
Serious Adverse Events (participants affected / at risk) | 0/409 | 0/417 | 0/326
Other Adverse Events (participants affected / at risk) | 0/409 | 0/417 | 0/326

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No